CLINICAL TRIAL: NCT06431256
Title: Phase 3, Multicenter, 3-Week Fixed-dose, Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy, Safety and PK Study of Evening Dosed Methylphenidate Hydrochloride ER Capsules (HLD200) in Children Aged 4-5 Years With ADHD
Brief Title: Efficacy, Safety & Pharmacokinetic (PK) Study of HLD200 in Children Aged 4-5 Years With ADHD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA release from this PMR study due to their required class-labeling, with a limitation of use for all ER stimulants in pediatric patients under 6 years of age, based on results from studies with other ER stimulants in this age group.
Sponsor: Ironshore Pharmaceuticals and Development, Inc (Other)
Collaborators: Collegium Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLD200-112
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo Comparator (Placebo Comparator): Matching placebo to HLD200 20 mg capsule (×2) for 3 weeks (prescribed at Visits 2, 3, and 4)
  Interventions: Drug: Placebo HLD200 capsules
- HLD200 20 mg (Experimental): HLD200 20 mg placebo capsule (×1) and HLD200 20 mg active capsule (×1) for 3 weeks (prescribed at Visits 2, 3, and 4)
  Interventions: Drug: HLD200 methylphenidate hydrochloride capsules
- HLD200 40 mg (Experimental): HLD200 20 mg placebo capsule (×1) and HLD200 20 mg active capsule (×1) for the first week (prescribed at Visit 2), with up-titration for the final 2 weeks to HLD200 20 mg active capsules (×2) (prescribed at Visits 3 and 4)
  Interventions: Drug: HLD200 methylphenidate hydrochloride capsules

INTERVENTIONS:
Drug: HLD200 methylphenidate hydrochloride capsules — Doses: 20mg capsules
  Other Names: methylphenidate
  Arms: HLD200 20 mg; HLD200 40 mg
Drug: Placebo HLD200 capsules — Doses: 20mg capsules
  Other Names: placebo
  Arms: Placebo Comparator

SUMMARY:
This study will evaluate the efficacy, safety and pharmacokinetics of HLD200 (20 mg and 40 mg) in children aged 4 to 5 years with ADHD.

DETAILED DESCRIPTION:
This is a multicenter, 3 week fixed dose, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy, safety and pharmacokinetics of HLD200 (20 mg and 40 mg) in children aged 4 to 5 years with ADHD.

Participants will be screened for eligibility for up to 4 weeks. Eligible participants will be treated with study medication for 3 weeks followed by a 2 week safety follow-up following the end of study treatment. The total duration of the study is up to 9 weeks. A single pharmacokinetic (PK) sample will be taken from each participant, in a prespecified PK sampling window at visit 5, for population PK analysis.

A total of 168 participants (56 per treatment arm) will be randomized at Visit 2.

ELIGIBILITY:
Inclusion Criteria:

1. The subject's assigned caregiver must be able to read, write, and/or understand at a level sufficient to provide informed consent and will provide this written consent (and subject will provide assent, if required by the IRB) before any study-specific activity is performed.
2. Subjects must be male or female children 4 to 5 years of age at the time of consent and assent (if applicable).
3. Subjects must have a diagnosis of ADHD as defined by the DSM-5 criteria with confirmation using the Mini - International Neuropsychiatric Interview for Children and Adolescents (MINI KID).
4. All subjects must have an ADHD-RS-IV Preschool Version Parent Total Score of ≥28 for boys or ≥24 for girls at Baseline (Visit 2). In addition, subjects not receiving pharmacotherapy for ADHD at time of consent must have an ADHD-RS-IV Preschool Version Parent Total Score of ≥28 for boys or ≥24 for girls at Screening; if the ADHD-RS-IV total score at Screening differs from the score at Baseline (Visit 2) by greater than 20% for these subjects (i.e., subjects who are not receiving ADHD pharmacotherapy at time of consent), the Investigator must investigate the reasons for the difference in score and determine whether the subject is an appropriate candidate to participate in the study.
5. Subjects not receiving pharmacotherapy for ADHD at time of consent must have a Clinical Global Impression - Severity (CGI-S) score ≥4 at Screening. All subjects must have a CGI-S score of ≥4 at Baseline (Visit 2).
6. Subjects must have a Peabody Picture Vocabulary Test 4 (PPVT-4) Standard Score ≥70 at Screening.
7. Subject has undergone an adequate course of nonpharmacologic treatment or has a severe enough condition in the opinion of the Investigator to consider enrollment without undergoing prior nonpharmacological treatment.
8. Subject's weight at Screening is between the 5th and 95th percentiles and subject's height at Screening is ≥ 5th percentile according to the Centers for Disease Control and Prevention growth charts by age and sex.
9. Subject must have a resting pulse less than 127 bpm, systolic and diastolic blood pressure below the 95th percentile for age, gender and height according to the 2017 American Academy of Pediatrics guidelines, based on the average of 3 measurements 2 to 5 minutes apart at Visit 1 and Visit 2 (only a single measurement is required at Visit 2 unless an elevated excursion is noted which requires the averaged value of triplicate measurements). If a subject's height is above the 95th percentile, the subject must meet the systolic and diastolic blood pressure criteria for the 95th percentile height.
10. Subject must be considered clinically appropriate for treatment with HLD200.
11. Subject must be in general good health based upon medical history, physical examination, clinical laboratory examinations, vital signs, and 12-lead electrocardiogram (ECG).
12. Subject and the subject's assigned caregiver are willing and able to participate in all study assessments and procedures, as applicable, and to follow all study requirements (including compliance with study drug), as described in the informed consent form.

Exclusion Criteria:

1. History of, or current, medical or psychiatric condition, including gastrointestinal disorders (e.g., surgery, malabsorption syndrome, and other similar conditions), open-angle glaucoma, abnormally increased intraocular pressure (IOP), or laboratory result that, in the opinion of the Investigator, unfavorably alters the risk-benefit of study participation, may jeopardize subject safety, or may interfere with the satisfactory completion of the study and study related procedures.
2. Serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, severe hypertension, untreated thyroid disease, peripheral vasculopathy, known structural cardiac disorders, serious cardiac conditions, serious arrhythmias, known family history of sudden death, or other cardiac problems that may place the subject at increased vulnerability to the sympathomimetic effects of a stimulant drug.
3. History of, or current, seizure disorder (except febrile seizures prior to age 4 and with last occurrence at least 1 year prior to study participation) or intellectual disability of mild severity or greater (DSM-5 criteria).
4. Past or current diagnosis of psychosis, bipolar I or II disorder, major depressive disorder, eating disorder, conduct disorder, obsessive-compulsive disorder, autism spectrum disorder, Tourette's Syndrome or other tic disorders, disruptive mood dysregulation disorder, or confirmed genetic disorder with cognitive and/or behavioral disturbances. Subjects with oppositional defiant disorder (ODD) or anxiety disorder (e.g., separation anxiety disorder simple phobia disorder) are permitted to enroll in the study provided these diagnoses are not the primary focus of treatment, and, in the opinion of the Investigator, are not anticipated to interfere with study assessments or procedures.
5. Subject is currently considered at risk of suicide in the opinion of the Investigator, or has previously made a suicide attempt, or has a history of, or is currently demonstrating active suicidal ideation or behavior, as determined by the C-SSRS at Screening and/or Baseline (Visit 2).
6. History of severe allergic reaction or intolerance to methylphenidate hydrochloride (MPH).
7. Alanine aminotransferase, aspartate aminotransferase, total bilirubin, or creatinine greater than 1.5 times the upper limit of normal. Elevated bilirubin due to Gilbert's syndrome is not exclusionary.
8. Use of ADHD stimulant medication within 72 hours (3 days) prior to Baseline (Visit 2); clonidine and guanfacine within 5 days prior to Baseline (Visit 2); psychotropic medications, including antidepressants (including MAOIs), mood stabilizers, and antipsychotics, within 14 days prior to Baseline (Visit 2); other prescription medications (including atomoxetine, excluding allowed medications) within 7 days prior to Baseline (Visit 2); and nonprescription/over-the-counter medications (excluding allowed medications) or herbal medications within the 3 days prior to Baseline (Visit 2). Medications not covered in allowed medications or prohibited medications must be cleared by the Medical Monitor prior to randomizing the subject.
9. Participation in a clinical trial with an investigational drug within the 30 days prior to Baseline (Visit 2).
10. Initiation of non-pharmacological treatment within 30 days prior to Baseline (Visit 2) or expected to initiate new non-pharmacological treatment during the study.
11. Use of any other medications that might confound the results of the study or increase risk to the subject.
12. In the opinion of the Investigator, the subject is well-controlled on his/her current ADHD medication with acceptable tolerability.
13. Subject has a sibling or step-sibling that is concurrently participating in this study or who has previously participated in this study.
14. Subject or caregiver is a participating Investigator, Sub-investigator, study coordinator, or employee of a participating Investigator, or is an immediate family member of the aforementioned.
15. Any factor, which in the opinion of the Investigator would jeopardize the evaluation or safety or be associated with poor adherence to the protocol.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Change in ADHD Rating Scale-IV (ADHD RS IV) Preschool Version | Day 1 (Baseline), Day 8, Day 15, Day 22
  The ADHD RS-IV Preschool Version measures the behaviors of children with ADHD and provides examples appropriate for the developmental level of preschool children. It is an 18-item questionnaire that requires the respondent to rate the frequency of occurrence of ADHD symptoms (as defined by DSM-IV-TR criteria) using a 4-point scale from 0 (rarely or never) to 3 (very often), with the total score ranging from 0 to 54; a decrease in score indicates an improvement in ADHD symptomology.

SECONDARY OUTCOMES:
Change in Clinical Global Impression - Severity (CGI-S) | Day 1 (Baseline), Day 8, Day 15, Day 22
  The investigator, or qualified designee, will rate the severity of a subject's condition on a 7-point scale ranging from 1 (normal) to 7 (among the most extremely ill subjects).
PK parameter: area under the plasma concentration-time curve (AUC) at steady-state (AUCss) | Day 22
  The PK of MPH will be determined using a single plasma sample collected at the end of treatment (Visit 5). Subjects will be randomly assigned to 1 of 4 PK sampling time points (11 hours, 14 hours, 18 hours, or 24 hours post-dose) for this single sample collection at Visit 5. The AUCss will be calculated based on the population PK model's individual predicted concentrations.
PK parameter: maximum plasma concentration (Cmax) | Day 22
  The PK of MPH will be determined using a single plasma sample collected at the end of treatment (Visit 5). Subjects will be randomly assigned to 1 of 4 PK sampling time points (11 hours, 14 hours, 18 hours, or 24 hours post-dose) for this single sample collection at Visit 5. The Cmax will be calculated based on the population PK model's individual predicted concentrations.
PK parameter: time to maximum plasma concentration (Tmax) | Day 22
  The PK of MPH will be determined using a single plasma sample collected at the end of treatment (Visit 5). Subjects will be randomly assigned to 1 of 4 PK sampling time points (11 hours, 14 hours, 18 hours, or 24 hours post-dose) for this single sample collection at Visit 5. The Tmax will be calculated based on the population PK model's individual predicted concentrations.
PK parameter: terminal elimination rate constant (λz) | Day 22
  The PK of MPH will be determined using a single plasma sample collected at the end of treatment (Visit 5). Subjects will be randomly assigned to 1 of 4 PK sampling time points (11 hours, 14 hours, 18 hours, or 24 hours post-dose) for this single sample collection at Visit 5. The λz will be calculated based on the population PK model's individual predicted concentrations.
PK terminal elimination half-life (t1/2) | Day 22
  The PK of MPH will be determined using a single plasma sample collected at the end of treatment (Visit 5). Subjects will be randomly assigned to 1 of 4 PK sampling time points (11 hours, 14 hours, 18 hours, or 24 hours post-dose) for this single sample collection at Visit 5. The t1/2 will be calculated based on the population PK model's individual predicted concentrations.
treatment-emergent adverse events (TEAEs) | Up to 5 weeks
  A TEAE is any newly occurring adverse event since the initiation of study drug treatment or any adverse event already present at the initiation of study drug treatment that worsens in either intensity or frequency during or after exposure to study drug treatment.
  Any clinically significant abnormal changes to ECG assessments, vital signs, clinical lab results, physical examinations, or sleep disturbance, or any suicidality during the trial, will be recorded as adverse events (unless they are signs/symptoms of a diagnosis already recorded as an AE).

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Harmonex, Inc., Dothan, Alabama
  - Advanced Research Center, Inc., Anaheim, California
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - South Florida Research, Miami Springs, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - DelRicht Research, New Orleans, Louisiana
  - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Vector Clinical Trials, Las Vegas, Nevada
  - University of Cincinnati Health, Cincinnati, Ohio
  - Coastal Pediatric Research, Summerville, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee